CLINICAL TRIAL: NCT00043979
Title: Pilot Study of Allogeneic/Syngeneic Blood Stem Cell Transplantation in Patients With High-Risk and Recurrent Pediatric Sarcomas
Brief Title: Stem Cell Transplantation in Patients With High-Risk and Recurrent Pediatric Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Terry Fry, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020259; 02-C-0259; NCT00047372 (obsolete NCT alias)
Record Dates: First submitted 2002-08-15; First posted 2002-08-16 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Sarcoma
Keywords: Ewing's Sarcoma; Rhabdomyosarcoma; Desmoplastic Small Round Cell Tumor; Sarcoma; Ewing Sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Desmoplastic Small Round Cell Tumor | interventions — Fluorodeoxyglucose F18; Cyclophosphamide; Cyclosporine; Doxorubicin; Etoposide; fludarabine phosphate; Melphalan; Prednisone; Sirolimus; Tacrolimus; Vincristine; Peripheral Blood Stem Cell Transplantation; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- Sibling Donors (Experimental): Donors (n = 30) were matched first degree relatives who were eligible to donate peripheral blood stem cells.
  Interventions: Drug: Filgrastim; Procedure: Peripheral Blood Stem Cell donation
- Arm 2 - Recipients (Experimental): Recipients (n=30) were enrolled to receive peripheral blood stem cells (PBSC) and receive either cyclosporine or tacrolimus and sirolimus for graft versus host disease (GVHD) prophylaxis.
  Interventions: Drug: F-18 Fluorodeoxyglucose; Biological: therapeutic allogeneic lymphocytes; Drug: cyclophosphamide; Drug: cyclosporine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: fludarabine phosphate; Drug: melphalan; Drug: prednisone; Drug: sirolimus; Drug: tacrolimus; Drug: vincristine sulfate; Procedure: peripheral blood stem cell transplantation; Drug: Filgrastim

INTERVENTIONS:
Drug: F-18 Fluorodeoxyglucose
  Other Names: FDG
  Arms: Arm 2 - Recipients
Biological: therapeutic allogeneic lymphocytes — Lymphocyte cells are collected from a healthy donor by apheresis and infused into the patient with a central venous catheter.
  Arms: Arm 2 - Recipients
Drug: cyclophosphamide — Induction - 750 mg/m^2 intravenous (IV) infusion over 30 minutes x 1 dose. Day 5.
  Transplant - 1200 mg/m^2 per day IV infusion over 2 hours daily for 4 days; days -6, -5, -4, -3.
  Other Names: Cytoxan
  Arms: Arm 2 - Recipients
Drug: cyclosporine — 6 mg/kg per dose orally every other day (no day 9 dose).
  Other Names: Sandimmune
  Arms: Arm 2 - Recipients
Drug: doxorubicin hydrochloride — Induction - 10 mg/m^2 per day continuous intravenous (IV) infusion over 24 hours daily for 4 days. Days 1, 2, 3, 4.
  Other Names: Adriamycin
  Arms: Arm 2 - Recipients
Drug: etoposide — 50 mg/m^2 per day continuous intravenous (IV) infusion over 24 hours daily for 4 days. Days 1, 2, 3, 4.
  Other Names: Vepesid
  Arms: Arm 2 - Recipients
Drug: fludarabine phosphate — Induction - 25 mg/m^2 per day intravenous (IV) infusion over 30 minutes daily for 3 days. Days 1, 2, 3.
  Transplant - 30 mg/m^2 per day IV infusion over 30 minutes daily for 4 days; days -6, -5, -4, -3.
  Other Names: Fludara
  Arms: Arm 2 - Recipients
Drug: melphalan — Transplant - 100 mg/m^2 per day intravenous (IV) infusion over 15 minutes for 1 day; day -2.
  Other Names: Alkeran
  Arms: Arm 2 - Recipients
Drug: prednisone — Induction - 60 mg/m^2 per day in 2-4 divided doses by mouth daily for 5 days; days 1, 2, 3, 4, 5.
  Other Names: Deltasone
  Arms: Arm 2 - Recipients
Drug: sirolimus — Initiated on day +3. Patients >40kg, the initial dose will be 2 mg every 24 hours orally. Patients <40 kg, the initial dose will be 1 mg/m^2.
  Other Names: Rapamune
  Arms: Arm 2 - Recipients
Drug: tacrolimus — Day -1 at least 24 hours before the stem cell infusion at a dose of 0.03 mg/kg/day as a continuous infusion. Twelve hours later oral dose initiated at a dose of 0.1-0.15 mg/kg/day in two divided doses every 12 hours.
  Other Names: Prograf
  Arms: Arm 2 - Recipients
Drug: vincristine sulfate — Induction - 0.4 mg/m^2 per day continuous intravenous (IV) infusion over 24 hours daily for 4 days; 1, 2, 3, 4.
  Other Names: Oncovin
  Arms: Arm 2 - Recipients
Procedure: peripheral blood stem cell transplantation — Stem cells from a healthy donor are collected and transplanted into the patient using a central venous catheter.
  Other Names: PBSCT
  Arms: Arm 2 - Recipients
Drug: Filgrastim
Procedure: Peripheral Blood Stem Cell donation
  Arms: Arm 1- Sibling Donors

SUMMARY:
This study will examine the safety and effectiveness of stem cell transplantation for treating patients with sarcomas (tumors of the bone, nerves, or soft tissue). Stem cells are immature cells in the bone marrow and blood stream that develop into blood cells. Stem cells transplanted from a healthy donor travel to the patient's bone marrow and begin producing normal cells. In patients with certain cancers, such as leukemia and lymphoma, the donor's immune cells attack the patient's cancer cells in what is called a "graft-versus-tumor" effect, contributing to cure of the disease. This study will determine whether this treatment can be used successfully to treat patients with sarcomas.

Patients between 4 and 35 years of age with a sarcoma that has spread from the primary site or cannot be removed surgically, and for whom effective treatment is not available, may be eligible for this study. Candidates must have been diagnosed by the age of 30 at the time of enrollment. They must have a matched donor (usually a sibling). Participants undergo the following procedures:

Donors: Stem cells are collected from the donor. To do this, the hormone granulocyte colony stimulating factor (G-CSF) is injected under the skin for several days to move stem cells out of the bone marrow into the bloodstream. Then, the cells are collected by apheresis. In this procedure the blood is drawn through a needle placed in one arm and pumped into a machine where the stem cells are separated out and removed. The rest of the blood is returned to the donor through a needle in the other arm.

Patients: For patients who do not already have a central venous catheter (plastic tube), one is placed into a major vein. This tube can stay in the body the entire treatment period for giving medications, transfusing blood, , withdrawing blood samples, and delivering the donated stem cells. Before the transplant procedure, patients receive from one to three cycles of "induction" chemotherapy, with each cycle consisting of 5 days of fludarabine, cyclophosphamide, etoposide, doxorubicin, vincristine, and prednisone followed by at least a 17-day rest period. All the drugs are infused through the catheter except prednisone, which is taken by mouth. After the induction therapy, the patient is admitted to the hospital for 5 days of chemotherapy with high doses of cyclophosphamide, melphalan, and fludarabine. Two days later, the stem cells are infused. The anticipated hospital stay is about 3 weeks, but may be longer if complications arise. Patients are discharged when their white cell count is near normal, they have no fever or infection, they can take sufficient food and fluids by mouth, and they have no signs of serious graft-versus-host disease (GVHD)-a condition in which the donor's cells "see" the patient's cells as foreign and mount an immune response against them.

After hospital discharge, patients are followed in the clinic at least once or twice weekly for a medical history, physical exam, and blood tests for 100 days. They receive medications to prevent infection and GVHD and, if needed, blood transfusions. If GVHD has not developed by about 120 days post transplant, patients receive additional white cells to boost the immune response. After 100 days, follow-up visits may be less frequent. Follow-up continues for at least 5 years. During the course of the study, patients undergo repeated medical evaluations, including blood tests and radiology studies, to check on the cancer and on any treatment side effects. On four occasions, white blood cells may be collected through apheresis to see if immune responses can be generated against the sarcomas treated in this study. Positron emission tomography (PET) scans may be done on five occasions. This test uses a radioactive material to produce images useful in detecting primary tumors and cancer that has spread.

DETAILED DESCRIPTION:
Background:

* Treatment of pediatric sarcomas has enjoyed progress in the past 25 years for patients with localized, chemosensitive disease and prognostic factors are now available to identify subsets of patients who have very dismal prognoses; patients with primary metastatic disease, especially those with bone and bone marrow metastases.
* Patients with primary chemoresistant disease and early recurrence also have very poor prognoses and lack suitable treatment options. For these patients, it is critical that alternative approaches to cytotoxic chemotherapy be identified.
* Basic laboratory studies have shown that Ewing's sarcoma is susceptible to immune mediated mechanisms of cytolysis in vitro. Interestingly, for Ewing's sarcoma this appears to be true for both chemosensitive and chemoresistant cell lines.
* Recent progress in the field of bone marrow transplantation has identified approaches that can reproducibly induce allogeneic peripheral blood stem cell engraftment in adults with hematologic malignancies. In some cases, this same approach has shown beneficial effects for patients with solid tumors as a result of the development of allogeneic, immune-mediated graft versus tumor effects.

Objectives:

* To determine if the transplantation of human leukocyte antigen (HLA) matched, peripheral blood stem cells can result in full donor engraftment (greater than 95 percent by day 100) in patients with high risk-pediatric sarcomas.
* To identify and characterize the toxicities of HLA-matched peripheral blood stem cell transplant (PBSCT) in patients with high-risk pediatric sarcomas. In particular we will identify the incidence of graft versus host disease (GVHD) and the pace of immune reconstitution in this population.
* To determine if allogeneic graft-versus-tumor responses following allogeneic PBSCT can induce clinically significant anti-tumor effects as measured by radiographic evidence of antitumor responses following PBSCT in patients with measurable disease and improved clinical outcome compared to historical controls in this patient population with a universally poor outcome.

Eligibility:

* Patients, age of greater than 4 years at enrollment to less than 30 years at diagnosis and age less than 35 at enrollment, with ultra-high risk Ewing's sarcoma family of tumors, desmoplastic small round cell tumor or alveolar rhabdomyosarcoma.
* Patients must have completed standard front-line therapy and salvage therapy.
* Patient must have the availability of a 5 or 6 antigen HLA-matched first-degree relative donor or a genotypically identical twin.
* Patients must have adequate cardiac, pulmonary, renal, liver, and marrow function.

Design:

-Donor will be prepared for peripheral blood stem cell harvest with Filgrastim mobilization, 10 microg/kg per day subcutaneous (SQ) for 5-7 days until they have stem cell collected by apheresis. The stem cells will then be cryopreserved.

Patients will receive 1 to 3 21 day cycles of Fludarabine-EPOCH induction chemotherapy. The preparative regimen will consist of cyclophosphamide, fludarabine and melphalan followed by stem cell infusion. GVHD prophylaxis will consist of sirolimus and tacrolimus.

ELIGIBILITY:
* INCLUSION CRITERIA: PATIENT

The following diagnoses will be considered:

1. Patients with Ewing's sarcoma family of tumors, or alveolar

   rhabdomyosarcoma in one of the following categories:
   * Patients who present at the time of initial diagnosis with bone or bone marrow metastases may be enrolled after completion of standard front-line therapy. Standard front line therapy for alveolar rhabdomyosarcoma should include vincristine and cyclophosphamide, plus actinomycin D and/or adriamycin. For patients with Ewing's sarcoma, standard front line therapy should include vincristine, cyclophosphamide, adriamycin, ifosfamide and etoposide.
   * Patients with recurrence of tumor at any site less than one year after completing standard front-line therapy or with a second or subsequent recurrence at any time after completing standard front-line therapy.
   * Patients with progression or persistence of disease while receiving standard front-line chemotherapy who cannot achieve a complete response (CR) with local treatment modalities.
2. The following patients with desmoplastic small round cell tumor are eligible after receiving front line standard therapy, which is defined as a regimen containing at least vincristine, cyclophosphamide, and adriamycin:

   * unresectable disease
   * metastatic tumor (abdominal and extra-abdominal disease)
   * progressive or persistent while receiving standard therapy
   * recurrence within one year of completing therapy

     * Patients without evaluable tumor at the time of enrollment are eligible
     * Patients who have previously received high-dose chemotherapy with autologous stem cell rescue are eligible for this trial.
     * Patient age 5-35 at enrollment.
     * Availability of a 5 or 6 antigen human leukocyte antigen (HLA)-matched first-degree relative donor (single HLA-A or B mismatch allowed). Genotypically identical twins may serve as stem cell donors. Genotypic identity must be confirmed by restrictive fragment length polymorphism (RFLP) analysis.
     * Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 or, for children less than or equal 10 years of age, Lansky greater than or equal 60
     * Cardiac function: Left ventricular ejection fraction greater than or equal to 45% by multi-gated acquisition scan (MUGA), fractional shortening greater than or equal 28% by echocardiogram (ECHO) or left ventricular ejection fraction greater than or equal 55% by ECHO.
     * Pulmonary function: carbon monoxide diffusing capacity (DLCO) greater than or equal to 50% of the expected value corrected for alveolar volume.
     * Renal function: Age-adjusted normal serum creatinine according to the following table or a creatinine clearance greater than or equal to 60 ml/min/1.73 m^2. Age (years) Maximum serum creatinine (mg/dl) less than or equal to 5 0.8 greater than 5, less than or equal to 10 1.0 greater than 10, less than or equal to15 1.2, greater than 15 1.5
     * Liver function: Serum total bilirubin less than 2 mg/dl, serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 times upper limit of normal.
     * Marrow function: absolute neutrophil count (ANC) must be greater than 750/mm^3 (unless due to underlying disease in which case there is no grade restriction), platelet count must be greater than or equal to 75,000/mm^3 (not achieved by transfusion) unless due to underlying disease in which case there is no grade restriction). Lymphopenia, cluster of differentiation 4 (CD4) lymphopenia, leukopenia, and anemia will not render patients ineligible.
     * Ability to give informed consent. For patients less than18 years of age their legal guardian must give informed consent. Pediatric patients will be included in age appropriate discussion in order to obtain verbal assent.
     * Durable power of attorney form completed (patients greater than or equal to18 years of age only).

INCLUSION CRITERIA: DONOR

* Weight greater than or equal 15 kilograms.
* First degree relative with genotypic identity at 5 or 6 HLA loci (single HLAA or B locus mismatch allowed). Genotypically identical twins may serve as stem cell donors. Genotypic identity must be confirmed by RFLP analysis.
* For donors less than 18 years of age, he/she must be the oldest suitable donor, their legal guardian must give informed consent, the donor must give verbal assent, and he/she must be cleared by social work and a mental health specialist to participate.
* For donors greater than or equal to 18 years of age, ability to give informed consent.
* Adequate peripheral venous access for apheresis or consent to use a temporary central venous catheter for apheresis.
* Donor selection criteria will be in accordance with National Institutes of Health (NIH)/Clinical Center (CC) Department of Transfusion Medicine Standards.

EXCLUSION CRITERIA: PATIENT

* Uncontrolled fungal infection.
* History of untreated CNS tumor involvement. Extradural masses which have not invaded the brain parenchyma (as is commonly observed in Ewing's sarcoma family of tumors) or parameningeal tumors (as is commonly observed in rhabdomyosarcoma) without evidence for leptomeningeal spread will not render the patient ineligible. Patients with previous central nervous system (CNS) tumor involvement that has been treated and has been stable for at least 6 weeks are eligible.
* Lactating or pregnant females.
* Human immunodeficiency virus (HIV) positive (due to unacceptable risk following allogeneic transplantation).
* Hepatitis B surface antigen (HBsAg) positive or hepatitis C antibody positive with elevated liver transaminases. All patients with chronic active hepatitis (including those on treatment) are ineligible.
* High risk of inability to comply with transplant protocol, or inability to give appropriate informed consent in the estimation of the principal investigator (PI), social work, or the stem cell transplant team.
* Fanconi Anemia

EXCLUSION CRITERIA: DONOR

* History of medical illness which poses a risk to donation in the estimation of the PI or the Department of Transfusion Medicine physician including, but not limited to stroke, hypertension that is not controlled with medication, or heart disease. Individuals with symptomatic angina or a history of coronary bypass grafting or angioplasty will not be eligible.
* History of congenital hematologic, immunologic, oncologic or metabolic disorder, which poses a prohibitive risk to the recipient in the estimation of the PI.
* Anemia (Hb less than 11 gm/dl) or thrombocytopenia (platelets less than 100,000/micro l).
* Lactating or pregnant females. Donors of childbearing potential must use an effective method of contraception during the time they are receiving growth colony stimulating factor (G-CSF). The effects of cytokine administration on a fetus are unknown and may be potentially harmful. The effects upon breast milk are also unknown and may potentially be harmful to the infant.
* Human immunodeficiency virus (HIV)-positive, hepatitis B surface antigen (HBsAg) positive or hepatitis C antibody positive. Donors are providing an allogeneic blood product and there is the potential risk of transmitting these viral illnesses to the recipient.
* High risk of inability to comply with transplant protocol.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2002-09-19 (Actual); Primary Completion 2009-05-01 (Actual); Study Completion 2011-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Fry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunst J, Sauer R, Burgers JM, Hawliczek R, Kurten R, Winkelmann W, Salzer-Kuntschik M, Muschenich M, Jurgens H. Radiation therapy as local treatment in Ewing's sarcoma. Results of the Cooperative Ewing's Sarcoma Studies CESS 81 and CESS 86. Cancer. 1991 Jun 1;67(11):2818-25. doi: 10.1002/1097-0142(19910601)67:113.0.co;2-y. PMID 2025847
- [Background] Demeocq F, Oberlin O, Benz-Lemoine E, Boilletot A, Gentet JC, Zucker JM, Behar C, Poutard P, Olive D, Brunat-Mentigny M, et al. Initial chemotherapy including ifosfamide in the management of Ewing's sarcoma: preliminary results. A protocol of the French Pediatric Oncology Society (SFOP). Cancer Chemother Pharmacol. 1989;24 Suppl 1:S45-7. doi: 10.1007/BF00253240. PMID 2667789
- [Background] Burdach S, Jurgens H, Peters C, Nurnberger W, Mauz-Korholz C, Korholz D, Paulussen M, Pape H, Dilloo D, Koscielniak E, et al. Myeloablative radiochemotherapy and hematopoietic stem-cell rescue in poor-prognosis Ewing's sarcoma. J Clin Oncol. 1993 Aug;11(8):1482-8. doi: 10.1200/JCO.1993.11.8.1482. PMID 8101562
- [Result] Baird K, Fry TJ, Steinberg SM, Bishop MR, Fowler DH, Delbrook CP, Humphrey JL, Rager A, Richards K, Wayne AS, Mackall CL. Reduced-intensity allogeneic stem cell transplantation in children and young adults with ultrahigh-risk pediatric sarcomas. Biol Blood Marrow Transplant. 2012 May;18(5):698-707. doi: 10.1016/j.bbmt.2011.08.020. Epub 2011 Sep 5. PMID 21896345
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0259.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sibling Donors: Donors (n = 30) were matched first degree relatives who were eligible to donate peripheral blood stem cells.In period 1 they donated cells.
- Recipients Cyclosporine GVHD Prophylaxis: In period 1 recipients received EPOCH-F/chemotherapy. In period 2 recipients received peripheral blood stem transplant.
  Post transplant recipients received cyclosporine for GVHD prophylaxis.
- Recipients Tacrolimus /Sirolimus Prophylaxis: In period 1 recipients received EPOCH-F/chemotherapy. In period 2 recipients received peripheral blood stem transplant.
  Post transplant recipients received tacrolimus & sirolimus for GVHD prophylaxis.
Period: Period 1
Arm/Group | Sibling Donors | Recipients Cyclosporine GVHD Prophylaxis | Recipients Tacrolimus /Sirolimus Prophylaxis
Started | 30 | 17 | 13
Completed | 23 | 13 | 10
Not Completed | 7 | 4 | 3
Not completed — recipient with progressive disease | 7 | 4 | 3
Period: Period 2
Arm/Group | Sibling Donors | Recipients Cyclosporine GVHD Prophylaxis | Recipients Tacrolimus /Sirolimus Prophylaxis
Started | 0 | 13 | 10
Completed | 0 | 13 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1-Sibling Donors: Donors (n=30) were matched first degree relatives who were eligible to donate peripheral blood stem cells.
- Arm 2-Recipients: Recipients (n=30) were enrolled to receive peripheral blood stem cells (PBSC) and receive either cyclosporine or tacrolimus and sirolimus for graft versus host disease (GVHD) prophylaxis.
- Total: Total of all reporting groups
Arm/Group | Arm 1-Sibling Donors | Arm 2-Recipients | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 14 | 31
  Between 18 and 65 years | 13 | 16 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.12 (10.9) | 19.98 (5.8) | 20.55 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 11 | 20 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Number of Prior Regimens of Participants that Received Stem Cell Transplant [Number; unit: regimens] — (c) Up-front regimen included autologous stem cell transplantation. Population: This baseline measure only applies to recipients.
  regimens
    Patient # 1: number analyzed (Participants) | 0 | 23 | 23
    Patient # 1 |  | 5 | 5
    Patient # 2: number analyzed (Participants) | 0 | 23 | 23
    Patient # 2 |  | 3 | 3
    Patient # 3: number analyzed (Participants) | 0 | 23 | 23
    Patient # 3 |  | 2 | 2
    Patient # 4: number analyzed (Participants) | 0 | 23 | 23
    Patient # 4 |  | 3 | 3
    Patient # 6: number analyzed (Participants) | 0 | 23 | 23
    Patient # 6 |  | 2 | 2
    Patient # 8: number analyzed (Participants) | 0 | 23 | 23
    Patient # 8 |  | 1 | 1
    Patient # 9: number analyzed (Participants) | 0 | 23 | 23
    Patient # 9 |  | 2 | 2
    Patient # 10: number analyzed (Participants) | 0 | 23 | 23
    Patient # 10 |  | 2 | 2
    Patient # 12: number analyzed (Participants) | 0 | 23 | 23
    Patient # 12 |  | 2 | 2
    Patient # 13: number analyzed (Participants) | 0 | 23 | 23
    Patient # 13 |  | 3 | 3
    Patient # 14: number analyzed (Participants) | 0 | 23 | 23
    Patient # 14 |  | 1 | 1
    Patient # 15: number analyzed (Participants) | 0 | 23 | 23
    Patient # 15 |  | 2 | 2
    Patient # 17: number analyzed (Participants) | 0 | 23 | 23
    Patient # 17 |  | 2 | 2
    Patient # 18: number analyzed (Participants) | 0 | 23 | 23
    Patient # 18 |  | 2 | 2
    Patient # 20: number analyzed (Participants) | 0 | 23 | 23
    Patient # 20 |  | 3 | 3
    Patient # 21: number analyzed (Participants) | 0 | 23 | 23
    Patient # 21 |  | 1 | 1
    Patient # 22: number analyzed (Participants) | 0 | 23 | 23
    Patient # 22 |  | 1 | 1
    Patient # 24: number analyzed (Participants) | 0 | 23 | 23
    Patient # 24 |  | 2 | 2
    Patient # 25: number analyzed (Participants) | 0 | 23 | 23
    Patient # 25 |  | 2 | 2
    Patient # 27: number analyzed (Participants) | 0 | 23 | 23
    Patient # 27 |  | 1 | 1
    Patient # 28 (c): number analyzed (Participants) | 0 | 23 | 23
    Patient # 28 (c) |  | 1 | 1
    Patient # 29: number analyzed (Participants) | 0 | 23 | 23
    Patient # 29 |  | 2 | 2
    Patient # 30: number analyzed (Participants) | 0 | 23 | 23
    Patient # 30 |  | 1 | 1
Number of Prior Regimens of Participants that Did Not Receive Stem Cell Transplant [Number; unit: regimens] — Population: This baseline measure applies to recipients only.
  regimens
    Patient # 5: number analyzed (Participants) | 0 | 7 | 7
    Patient # 5 |  | 2 | 2
    Patient # 7: number analyzed (Participants) | 0 | 7 | 7
    Patient # 7 |  | 1 | 1
    Patient # 11: number analyzed (Participants) | 0 | 7 | 7
    Patient # 11 |  | 3 | 3
    Patient # 16: number analyzed (Participants) | 0 | 7 | 7
    Patient # 16 |  | 2 | 2
    Patient # 19: number analyzed (Participants) | 0 | 7 | 7
    Patient # 19 |  | 2 | 2
    Patient # 23: number analyzed (Participants) | 0 | 7 | 7
    Patient # 23 |  | 4 | 4
    Patient # 26: number analyzed (Participants) | 0 | 7 | 7
    Patient # 26 |  | 3 | 3
Participants who Received Stem Cell Transplant Disease Status at Enrollment [Count of Participants; unit: Participants] — Population: This baseline measure applies to recipients only.
  Participants
    Progressive Disease (PD): number analyzed (Participants) | 0 | 23 | 23
    Progressive Disease (PD) |  | 18 | 18
    No Evidence of Disease (NED): number analyzed (Participants) | 0 | 23 | 23
    No Evidence of Disease (NED) |  | 4 | 4
    Stable Disease (SD): number analyzed (Participants) | 0 | 23 | 23
    Stable Disease (SD) |  | 1 | 1
Participants who Did Not Receive Stem Cell Transplant Disease Status(Progressive Disease)/Enrollment [Count of Participants; unit: Participants] — Population: This baseline measure applies to recipients only.
  Participants
    number analyzed (Participants) | 0 | 7 | 7
    (all) |  | 7 | 7
Disease Status at Hematopoietic Stem Cell Transplant [Count of Participants; unit: Participants] — This list includes the disease status of participants who received stem cell transplant. Population: This baseline measure applies to recipients only.
  Participants
    Partial Response (PR): number analyzed (Participants) | 0 | 23 | 23
    Partial Response (PR) |  | 4 | 4
    Stable Disease (SD): number analyzed (Participants) | 0 | 23 | 23
    Stable Disease (SD) |  | 9 | 9
    No Evidence of Disease (NED): number analyzed (Participants) | 0 | 23 | 23
    No Evidence of Disease (NED) |  | 4 | 4
    Progressive Disease (PD): number analyzed (Participants) | 0 | 23 | 23
    Progressive Disease (PD) |  | 3 | 3
    Complete Response (CR)/(NED): number analyzed (Participants) | 0 | 23 | 23
    Complete Response (CR)/(NED) |  | 3 | 3
Disease Status (Progressive Disease) at Hematopoietic Stem Cell Transplant [Count of Participants; unit: Participants] — This list includes the disease status of participants who did not receive stem cell transplant. Population: This baseline measure applies to recipients only.
  Participants
    number analyzed (Participants) | 0 | 7 | 7
    (all) |  | 7 | 7
Diagnosis (Participants that Received Stem Cell Transplant) [Count of Participants; unit: Participants] — aRMS indicates alveolar rhabdomyosarcoma; ESRT, Ewings sarcoma; DSRCT, desmoplastic small round cell tumor. Population: This baseline measure applies to recipients only.
  Participants
    aRMS: number analyzed (Participants) | 0 | 23 | 23
    aRMS |  | 7 | 7
    ESFT: number analyzed (Participants) | 0 | 23 | 23
    ESFT |  | 5 | 5
    DSRCT: number analyzed (Participants) | 0 | 23 | 23
    DSRCT |  | 11 | 11
Diagnosis (Participants that Did Not Receive Stem Cell Transplant) [Count of Participants; unit: Participants] — ESRT, Ewings sarcoma; DSRCT, desmoplastic small round cell tumor. Population: This baseline measure applies to recipients only.
  Participants
    ESFT: number analyzed (Participants) | 0 | 7 | 7
    ESFT |  | 6 | 6
    DSRCT: number analyzed (Participants) | 0 | 23 | 23
    DSRCT |  | 1 | 1
High-Risk Features (Participants that Received Stem Cell Transplant) [Count of Participants; unit: Participants] — B/BM indicates bone or bone marrow metastases; ER, early recurrence; MR, multiply recurrent; PP, primary progressive disease. Population: This baseline measure applies to recipients only.
  Participants
    MR: number analyzed (Participants) | 0 | 23 | 23
    MR |  | 6 | 6
    ER: number analyzed (Participants) | 0 | 23 | 23
    ER |  | 2 | 2
    ER, B/BM, MR: number analyzed (Participants) | 0 | 23 | 23
    ER, B/BM, MR |  | 1 | 1
    PP: number analyzed (Participants) | 0 | 23 | 23
    PP |  | 1 | 1
    B/BM: number analyzed (Participants) | 0 | 23 | 23
    B/BM |  | 7 | 7
    Metastatic: number analyzed (Participants) | 0 | 23 | 23
    Metastatic |  | 4 | 4
    PP/Metastatic: number analyzed (Participants) | 0 | 23 | 23
    PP/Metastatic |  | 1 | 1
    PP, B/BM: number analyzed (Participants) | 0 | 23 | 23
    PP, B/BM |  | 1 | 1
High-Risk Features (Participants that Did Not Receive Stem Cell Transplant) [Count of Participants; unit: Participants] — B/BM indicates bone or bone marrow metastases; ER, early recurrence; MR, multiply recurrent; PP, primary progressive disease. Population: This baseline measure applies to recipients only.
  Participants
    ER, B/BM: number analyzed (Participants) | 0 | 7 | 7
    ER, B/BM |  | 1 | 1
    PP, B/BM: number analyzed (Participants) | 0 | 7 | 7
    PP, B/BM |  | 1 | 1
    ER: number analyzed (Participants) | 0 | 7 | 7
    ER |  | 3 | 3
    PP: number analyzed (Participants) | 0 | 7 | 7
    PP |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment
Description: Engraftment is defined as rapid conversion to complete donor chimerism and is assessed by blood counts and chimerism, >95% donor engraftment at day 100 in >75% of patients.
Time Frame: 100 days
Population: E.g ...in >75% of patients, shown above is not a conclusion but refers to a hypothesis, the objective of the protocol.
  23 were analyzed because 7 donors were taken off study and stem cells not collected due to progressive disease of sibling.
Measure: Number; unit: Participants
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 23
Participants | 23

2. Primary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 16.5 months
Measure: Number; unit: Participants
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 30
Participants | 30

3. Secondary Outcome: Number of Participants With Acute and Chronic GVHD
Description: Acute GVHD as by Modified Glucksberg Criteria occurring before day 100. Chronic GVHD as per Seattle criteria occurring after day 100.
Time Frame: up to 5 years or death
Measure: Number; unit: participants
Arm/Group | Recipients -Cyclosporine GVHD Prophylaxis | Recipients -Tacrolimus/Sirolimus GVHD Prophylaxis
Number analyzed (Participants) | 13 | 10
participants
  acute GVHD | 12 | 5
  chronic GVHD | 12 | 5

4. Secondary Outcome: Median Time to Reach Absolute Neutrophil Count of 500/mm(3)
Description: Days for participants to achieve a neutrophil count of 500/mm(3).
Time Frame: up to 12 days
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 30
Days | 9 [8 to 12]

5. Secondary Outcome: Median Time to Reach a Platelet Count of 50,000/mm(3)
Description: Days for participants to achieve a platelet count of 50,000/mm(3).
Time Frame: up to 43 days
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 30
Days | 15 [10 to 43]

6. Secondary Outcome: Early Post Transplantation Relapse
Description: Participants who experienced recurrence or progression of disease following transplant.
Time Frame: up to 300 days
Population: One out of 23 participants did not have a recurrence, thus was excluded from analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 22
Days | 100 [28 to 300]

7. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival was based on the time from on-study date until progression or last follow-up.
Time Frame: up to 77 months
Population: 23 were analyzed because 7 donors were taken off study and stem cells not collected due to progressive disease of sibling.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 23
Months | 15.9 [2.2 to 77.0]

8. Secondary Outcome: Two Year Survival Rate for Patients Undergoing Allo-Hematopoietic Stem Cell Transplant
Description: Participants who are alive at two years following Allo-Hematopoietic Stem Cell Transplant.
Time Frame: 2 years
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 23
percentage of participants
  From date of enrollment | 39.1
  From date of transplantation | 34.8

9. Secondary Outcome: Number of Participants to Complete Conversion to >95% Donor Chimerism
Description: Participants who tolerated the transplantation regimen and accepted >95% of the donors blood, marrow, and/or tissue.
Time Frame: up to 30 days
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 23
Participants
  Day +14 | 23
  Day +28 | 23

10. Secondary Outcome: Cluster of Differentiation 4 (CD4) Reconstitution
Description: The median CD4 count with a range of 85-1565 (absolute count) was used to determine recovery and were considered recovered if in this range. The CD4 count was established by flow cytometry testing.
Time Frame: Day +28-42
Measure: Median (Full Range); unit: mm(3)
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 30
mm(3) | 284 [85 to 1042]

11. Secondary Outcome: Best Response Post-Hematopoietic Stem Cell Transplant EOCH (Etoposide, Vincristine, Cyclophosphamide, and Doxorubicin)
Description: Response is defined by the Response Evaluation Criteria in Solid Tumors (RECIST). RECIST criteria offer a simplified, conservative, extraction of imaging data for wide application in clinical trials. They presume that linear measures are an adequate substitute for 2-D (dimensional) methods and registers four response categories: Complete response (CR) is disappearance of all target lesions. Partial response (PR) is 30% increase in the sum of the longest diameter of target lesions. Progressive disease (PD) is 20% increase in the sum of the longest diameter of target lesions. Stable disease (SD) is small changes that do not meet above criteria. For the purposes of this study very good partial response ((VGPR) is >75% reduction in disease) was also employed.
Time Frame: up to 10 cycles of therapy or 280 days
Population: EPOCH-F (Etoposide, Vincristine, Prednisone, Cyclophosphamide, Doxorubicin, and Fludarabine) was modified to EOCH and administered to 12 patients for post-transplantation disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 12
Participants
  Complete Response (CR) | 2
  Progressive Disease (PD) | 4
  Partial Response (PR) | 4
  Very Good Partial Response (VGPR) | 2

12. Secondary Outcome: Median Survival From Date of Progression
Description: Median survival from date of progression is based on the time from on-study date until progression or last follow-up.
Time Frame: up to 77 months
Population: as for outcome 7
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 23
Months
  Participants who did not receive a transplant(n=7) | 3.3 [2.2 to 11.2]
  Participants who received a transplant (n=23) | 19.1 [5.6 to 77.0]
Statistical Analysis 1: Comparison: Arm 2-Recipients; Test type: Superiority or Other; p = .0003, Kaplan-Meier — 7 participants who did not receive a transplant compared with 21 participants transplanted

13. Other Pre Specified Outcome: Number of Participants Who Experienced Graft Versus Tumor Effect (GVT)
Description: GVT is defined as tumor response after day 42 post-transplantation without cytotoxic therapy.
Time Frame: up to day 100
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 23
Participants | 0

14. Other Pre Specified Outcome: Post-Hematopoietic Stem Cell Transplant (HSCT) Radiotherapy
Description: Site of radiotherapy (high energy radiation) and/or toxicity experienced by the participants post HSCT radiotherapy. Grading was preformed using the Modified Glucksberg Criteria.
Time Frame: up to 6 cycles or 168 days
Population: G1, grade 1; G2, grade 2; G3, grade 3; G4, grade 4; G5, grade 5. 23 were analyzed because 7 donors were taken off study and stem cells not collected due to progressive disease of sibling.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2-Recipients
Number analyzed (Participants) | 23
Participants
  Chest wall; G2 skin | 1
  Abdomen; G4 GI | 1
  Pancreas; G4 LFTs, G4 pancreatitis | 1
  Pleura, mediastinum; G4 LFTs, G2 mucositis | 1
  Chest wall; G4 skin, G3 mucositis | 1
  Spine, skull; G2 nausea+vomiting, G2 fatigue | 1
  Pelvis; G4 enteritis | 1
  Pulmonary (cyberknife) | 1
  Brain; B3 mucositis | 1
  Whole lung; G3 mucositis, G3 skin, G5 lung | 1
  L arm, R shoulder, B/L femur | 1

ADVERSE EVENTS:
Time Frame: 16.5 months
Arm/Group | Arm 2-Recipients
All-Cause Mortality (participants affected / at risk) | 29/30
Serious Adverse Events (participants affected / at risk) | 29/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2-Recipients (N=30)
Cardiac General: Hypotension (Cardiac disorders) | 1 (1)
Constitutional Symptoms: Fever (General disorders) | 1 (1) — (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Creatinine (Renal and urinary disorders) | 1 (1)
Death: Death not associated with CTCAE term: Disease progression NOS (General disorders) | 29 (29)
Gastrointestinal: Diarrhea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal:Mucositis/stomatitis (clinical exam)::oral cavity (Gastrointestinal disorders) | 1 (1)
GI, other (Gastrointestinal disorders) | 1 (1)
Infection with neutropenia (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1)
Infection: Febrile neutropenia (Infections and infestations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >=38.5 degrees C)
Intussception (Gastrointestinal disorders) | 1 (1)
Metabolic/Laboratory: Bilirubin, serum-high (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Metabolic/Laboratory: ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory: AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Mood alteration; suicide gesture (Nervous system disorders) | 1 (1)
Neurology: Mood alteration: anxiety (Nervous system disorders) | 1 (1)
Neurology: Seizure (Nervous system disorders) | 2 (2)
Pain - right chest wall (General disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pulmonary/Upper Respiratory: Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary - Other (pulmonary edema w/normal 02 sat) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory: Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/Upper Respiratory: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Radiation Recall Reaction (anterior chest) (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Thrombosis (Cardiac disorders) | 2 (2)
Vaginitis (Renal and urinary disorders) | 1 (1)
AST, high (Metabolism and nutrition disorders) | 1 (1)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 (3)
Pneumonitits/Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2-Recipients (N=30)
Abdominal cramping (Gastrointestinal disorders) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abscesses (crypt) (Gastrointestinal disorders) | 1 (1)
Acne breakout (Skin and subcutaneous tissue disorders) | 1 (1)
Adenopathy (Blood and lymphatic system disorders) | 1 (1)
Agitated mental status (Nervous system disorders) | 1 (1)
Albumin low (Hepatobiliary disorders) | 1 (1)
Alk. phosph. (Hepatobiliary disorders) | 1 (1)
Allergic rhinitis-rhinorrhea (Immune system disorders) | 1 (1)
Allergy/Immunology: Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Allergy/Immunology: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 18 (60)
Allergy/Immunology: Autoimmune reaction (Immune system disorders) | 1 (5)
Appetite decreased (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bacteremia (Blood and lymphatic system disorders) | 2 (2)
Bilious emesis (Gastrointestinal disorders) | 1 (1)
Bilious vomiting (Gastrointestinal disorders) | 1 (1)
Blood/Bone Marrow:Platelets (Blood and lymphatic system disorders) | 26 (375)
Blood/Bone Marrow:Hemoglobin (Blood and lymphatic system disorders) | 30 (393)
Blood/Bone Marrow:Leukocytes (total WBC) (Blood and lymphatic system disorders) | 27 (241)
Blood/Bone Marrow:Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 26 (235)
Blurred vision (Eye disorders) | 3 (3)
Bullous myringitis (Ear and labyrinth disorders) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Burns, radiation (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Arrhythmia: Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 7 (13)
Cardiac General: Hypertension (Cardiac disorders) | 7 (16)
Cardiac General:Hypotension (Cardiac disorders) | 9 (20)
Chills (General disorders) | 3 (3)
Compression of vena cava by tumor (Cardiac disorders) | 1 (1)
Congestion (Immune system disorders) | 3 (3)
Constitutional Symptoms - Other (pallor) (General disorders) | 1 (1)
Constitutional Symptoms: Fatigue (asthenia, lethargy, malaise) (General disorders) | 20 (43)
Constitutional Symptoms: Fever (General disorders) | 20 (55) — (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Constitutional Symptoms: Insomnia (General disorders) | 6 (11)
Constitutional Symptoms: Weight loss (General disorders) | 6 (11)
Creatinine (Renal and urinary disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 4 (4)
Dermatology/Skin: Pigmentation changes (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatology/Skin: Dermatology/Skin-Other (lip abrasion) (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin: Dermatology/Skin-Other (specify: verrucae) (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatology/Skin: Dry skin (Skin and subcutaneous tissue disorders) | 9 (29)
Dermatology/Skin: Rash/dermatitis associated with high dose chemotherapy or BMT studies (Skin and subcutaneous tissue disorders) | 1 (11)
Dermatology/Skin: Rash: acne (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatology/Skin: Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 6 (14)
Dermatology/Skin: Dermatology/Skin-Other (specify, keratosis pilaris) (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatology/Skin: Hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (10)
Dermatology/Skin: Nail changes (Skin and subcutaneous tissue disorders) | 2 (5)
Dermatology/Skin: Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (4)
Dermatology/Skin: Rash/desquamation (Skin and subcutaneous tissue disorders) | 15 (130)
Dermatology/Skin: Rash/desquamation associated with graft versus host disease (GVHD) (Skin and subcutaneous tissue disorders) | 5 (28) — for BMT studies, if specified in the protocol
Dermatology/Skin: Rash: dermatitis associated with radiation-select: radiation (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin: Striae (Skin and subcutaneous tissue disorders) | 1 (5)
Desquamation of palmar surface of hands, B/L (Skin and subcutaneous tissue disorders) | 1 (1)
Desquamation, vaginal (Skin and subcutaneous tissue disorders) | 1 (1)
Diaphoresis (General disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspareunia (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Dystonia (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3)
Ears-dry (Ear and labyrinth disorders) | 1 (1)
Edema, extremities (Blood and lymphatic system disorders) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (1)
Endocrine: Cushingoid appearance (Endocrine disorders) | 9 (29)
Epidermal abrasions (Skin and subcutaneous tissue disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema, palms of hands (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema - abdominal incision (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema - buccal mucosa (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema-face (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema - right great toe pus (Skin and subcutaneous tissue disorders) | 1 (1)
Erythemateous patchy rash - mild, primarily involving trunk but listed (back, chest, arms) (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis, chronic (Gastrointestinal disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eyes - dry bilateral (Eye disorders) | 1 (1)
Fibrosis lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fissure (General disorders) | 1 (1)
Flat effect (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Gastrointestinal: Anorexia (Gastrointestinal disorders) | 10 (16)
Gastrointestinal:Constipation (Gastrointestinal disorders) | 13 (24)
Gastrointestinal:Dental: periodontal disease (Gastrointestinal disorders) | 1 (5)
Gastrointestinal:Diarrhea (Gastrointestinal disorders) | 22 (74)
Gastrointestinal:Distention, bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Gastrointestinal:Flatulence (Gastrointestinal disorders) | 2 (3)
Gastrointestinal:Heartburn/Dyspepsia (Gastrointestinal disorders) | 5 (10)
Gastrointestinal:Hemorrhoids (Gastrointestinal disorders) | 2 (7)
Gastrointestinal:Mucositis/stomatitis (clinical exam)::oral cavity (Gastrointestinal disorders) | 9 (14)
Gastrointestinal:Mucositis/stomatitis (functional/symptomatic)::pharynx (Gastrointestinal disorders) | 2 (3)
Gastrointestinal:Nausea (Gastrointestinal disorders) | 21 (44)
GVHD (Gastrointestinal disorders) | 4 (12)
GVHD, GI (Gastrointestinal disorders) | 2 (2)
GVHD - cutaneous (Gastrointestinal disorders) | 1 (1)
GVHD, GI & skin & liver (Gastrointestinal disorders) | 2 (2)
GVHD, liver (Gastrointestinal disorders) | 1 (1)
GVHD: skin, liver, oral and vaginal mucosa (Gastrointestinal disorders) | 1 (1)
GVHD - skin, liver, oral buccal mucosa (Gastrointestinal disorders) | 1 (1)
Hallucination(s) (Nervous system disorders) | 2 (2)
Headache (General disorders) | 5 (6)
Headaches-intermittent (General disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhage, epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hemorrhage/Bleeding: Hemorrhage, pulmonary/upper respiratory-select (Respiratory, thoracic and mediastinal disorders) | 1 (2) — hemorrhage, pulmonary/upper respiratory - pleura
Hemorrhage/Bleeding: Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 4 (7)
Hemorrhage/Bleeding: Vagina (Reproductive system and breast disorders) | 1 (3)
Hepatic: Bilirubin associated with graft versus host disease (GVHD) for BMT studies, (Hepatobiliary disorders) | 4 (8) — if specified in the protocol
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoxia-Hypoxemic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased cavitary nodular infiltrate in left lower lobe (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infection-Other (Infections and infestations) | 3 (5)
Infection-Other (specify) tinea pedis, left foot (Infections and infestations) | 1 (1)
Infection - sexual/reproductive function - vulva (Infections and infestations) | 1 (1)
Infection w/neutropenia (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 4 (4)
Infection, C. diff & rota virus (Infections and infestations) | 1 (1)
Infection, CVL (Infections and infestations) | 1 (1)
Infection, influenza (w/o neutropenia) (Infections and infestations) | 1 (1)
Infection, musculo-skeletal, soft tissue (Infections and infestations) | 1 (1)
Infection: Febrile neutropenia (Infections and infestations) | 5 (5) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >=38.5 degrees C)
Infection: Infection (Infections and infestations) | 5 (5) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC<1.0x10e9/L): pulmonary/upper respiratory - lung (pneumonia)
Infection: Infection (documented clinically or microbiologically) (Infections and infestations) | 4 (5) — with Grade 3 or 4 neutrophils (ANC<1.0x10e9/L): skin (cellulites)
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: (Infections and infestations) | 1 (1) — pulmonary/upper respiratory, upper airway NOS
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: select - conjunctiva (Infections and infestations) | 4 (8)
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: skin (Infections and infestations) | 1 (1)
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: skin (cellulitis) (Infections and infestations) | 1 (1)
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: upper airway NOS (Infections and infestations) | 1 (1)
Infection-upper respiratory symptoms (Infections and infestations) | 1 (1)
Infiltrate (lung) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intermittent headache (General disorders) | 1 (1)
Itching (anal warts) (Gastrointestinal disorders) | 1 (1)
Joint soreness, intermittent (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness & pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Low energy level (General disorders) | 1 (1)
Low grade fever (General disorders) | 2 (2)
Lymphatics (Blood and lymphatic system disorders) | 1 (1)
Lymphatics: edema: limb (Blood and lymphatic system disorders) | 5 (8)
Lymphocytes (Blood and lymphatic system disorders) | 4 (4)
Macular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Macular rash on anterior and posterior chest (Skin and subcutaneous tissue disorders) | 1 (1)
Metabolic/Laboratory: Bilirubin, serum-high (hyperbilirubinemia) (Metabolism and nutrition disorders) | 21 (134)
Metabolic/Laboratory: Other (Urea nitrogen, low???) (Metabolism and nutrition disorders) | 8 (27)
Metabolic/Laboratory: Cholesterol, serum high (hypercholestremia) (Metabolism and nutrition disorders) | 6 (23)
Metabolic/Laboratory: AST, SGOT (serum glutamic oxaloacetic) (Metabolism and nutrition disorders) | 24 (253)
Metabolic/Laboratory: Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 24 (163)
Metabolic/Laboratory: Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 27 (408)
Metabolic/Laboratory: Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 8 (14)
Metabolic/Laboratory: Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 15 (43)
Metabolic/Laboratory: Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 22 (153)
Metabolic/Laboratory: Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 9 (14)
Metabolic/Laboratory: Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 25 (165)
Metabolic/Laboratory: Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 8 (36)
Mg, low (Metabolism and nutrition disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 1 (1)
Mild constipation (Gastrointestinal disorders) | 1 (1)
Mild cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mild nasal congestion (Immune system disorders) | 1 (1)
Mild neuropathy of right foot (Nervous system disorders) | 1 (1)
Mild tenderness in lumbosacral area (Musculoskeletal and connective tissue disorders) | 1 (1)
Molluscum rash to upper thighs B/L (Skin and subcutaneous tissue disorders) | 1 (1)
Mood alteration - anxiety (Nervous system disorders) | 3 (3)
Mood alteration-depression (Nervous system disorders) | 2 (2)
Muscle aches-back, hip, left neck, right lateral chest wall, right scapular (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/other-joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft tissue: joint-effusion (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal/Soft tissue: Muscle weakness, genralized or specific area (Musculoskeletal and connective tissue disorders) | 1 (1) — (not due to neuropathy) - select- extremity-lower
Musculoskeletal/Soft tissue: Fracture (Musculoskeletal and connective tissue disorders) | 2 (7)
Musculoskeletal/Soft tissue: Muscle weakness, generalized or specific area (not due to neuropathy): (Musculoskeletal and connective tissue disorders) | 2 (7) — Extremity-lower
Musculoskeletal/Soft tissue: Musculoskeletal/Soft tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (5) — (specify, radiation changes to pelvis)
Musculoskeletal/Soft tissue: Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 2 (6)
Myalgia-Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Neurology: Mood alteration: agitation (Nervous system disorders) | 2 (3)
Neurology: mood alteration: anxiety (Nervous system disorders) | 9 (21)
Neurology: mood alteration: depression (Nervous system disorders) | 12 (27)
Neurology: neuropathy: cranial - select neuropathy: CN XII motor- tongue (Nervous system disorders) | 1 (1)
Neurology: neuropathy: sensory (Nervous system disorders) | 7 (20)
Neurology: seizure (Nervous system disorders) | 2 (3)
Neurology: tremor (Nervous system disorders) | 9 (19)
Neuropathy (Nervous system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Ocular/Visual: dry eye syndrome (Eye disorders) | 2 (9)
Ocular/Visual: cataract (Eye disorders) | 1 (2)
Ocular/Visual: Ocular/Visual - Other (specify, erythema) (Eye disorders) | 1 (5)
Ocular/Visual: Vision-blurred vision (Eye disorders) | 2 (2)
Oral candidiasis (Gastrointestinal disorders) | 1 (3)
Oral pain, esophageal pain (Gastrointestinal disorders) | 1 (1)
Other, edema (Blood and lymphatic system disorders) | 1 (1)
Other, fluid overload (Blood and lymphatic system disorders) | 1 (1)
Other, sixth nerve palsy (Nervous system disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pain, head (General disorders) | 1 (1)
Pain mouth sore (Gastrointestinal disorders) | 1 (1)
Pain perianal (Gastrointestinal disorders) | 1 (1)
Pain thoracic (General disorders) | 1 (1)
Pain, abdominal (Gastrointestinal disorders) | 8 (9)
Pain, chest (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, extremities (throbbing) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Headache (Nervous system disorders) | 3 (3)
Pain, knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, left trapezius and shoulder area (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain, oral mucosa (Gastrointestinal disorders) | 1 (1)
Pain, ear (Ear and labyrinth disorders) | 1 (1)
Pain, musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, tenderness (chest) (Musculoskeletal and connective tissue disorders) | 1 (1)
pain/auditory/ear: external (Ear and labyrinth disorders) | 1 (1)
Coagulation: PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 28 (159)
Colitis (Gastrointestinal disorders) | 1 (1)
Pain/Gastrointestinal:dental/teeth/periodontal (Gastrointestinal disorders) | 1 (2)
Pain/Musculoskeletal:Back (Musculoskeletal and connective tissue disorders) | 8 (20)
Pain/Musculoskeletal:Extremity-limb (Musculoskeletal and connective tissue disorders) | 9 (26)
Pain/Musculoskeletal:Bone (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain/Musculoskeletal:Buttock (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain/Musculoskeletal:Neck (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain/Neurology:Head/Headache (Nervous system disorders) | 6 (12)
Pain/Ocular: eye (Eye disorders) | 1 (2)
Pain/Pulmonary/Upper Respiratory: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pain/Pulmonary/Upper Respiratory:Chest wall (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pain/Pulmonary/Upper Respiratory:Pleura (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain/Pulmonary/Upper Respiratory:Sinus (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pain:Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: pleuritic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain:vaginally (Reproductive system and breast disorders) | 1 (1)
Pain:Gastrointestinal: oral cavity (Gastrointestinal disorders) | 3 (8)
Papular rash hands (Skin and subcutaneous tissue disorders) | 1 (1)
Paronychia, hallux, B/L (Infections and infestations) | 1 (1)
Peeling-bilateral palms (Skin and subcutaneous tissue disorders) | 1 (1)
Pericardial fluid (Cardiac disorders) | 1 (1)
Poor appetite (Gastrointestinal disorders) | 3 (3)
Positive viral culture (Infections and infestations) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Psychotic episode (Psychiatric disorders) | 1 (1)
PT, prolonged (Blood and lymphatic system disorders) | 8 (8)
RBC transfusion (Blood and lymphatic system disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, other, tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sweating (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1)
Transfusion, platelet (Blood and lymphatic system disorders) | 2 (2)
Ulcer, duodenal (Gastrointestinal disorders) | 1 (1)
Ulcers near molars (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Uveitis, OU (Eye disorders) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
Vertigo (sensation) (Nervous system disorders) | 1 (1)
Visual hallucination (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (9)
Xeropthalmia (Eye disorders) | 1 (1)
Infection: Infection with normal ANC or Grade 1 or 2 neutrophils: Dermatology-Skin (Infections and infestations) | 1 (1)
Metabolic/Laboratory: Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 10 (26)
Pain: Musculoskeletal - Joint (Musculoskeletal and connective tissue disorders) | 7 (11)
Pain: NOS (General disorders) | 1 (2)
Pain: Pain: Auditory/Ear (Ear and labyrinth disorders) | 1 (1)
Pain-ankles & knees (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - back (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain - chest (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - left eye (Eye disorders) | 1 (1)
Pain - right eye (Eye disorders) | 1 (1)
Pain - scapular (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - skull (Musculoskeletal and connective tissue disorders) | 1 (1)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pansinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Patchy erythema, upper and lower extremities, palms and soles, B/L (Skin and subcutaneous tissue disorders) | 1 (1)
Perianal pain (Gastrointestinal disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Phosphatemia (Metabolism and nutrition disorders) | 2 (2)
Pigmentation changes (Skin and subcutaneous tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post-nasal drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Protein low (Metabolism and nutrition disorders) | 1 (1)
Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory: Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory: Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory: Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory: Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Radiation Dermatits (Skin and subcutaneous tissue disorders) | 2 (2)
Rash - erythematous, mild, lacy (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - trunk, arms, face, legs, sparing feet (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Acne) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (maculopapular) GVHD (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (port erythema) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, B/L LEs and UEs (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, erythematous (GVHD) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, palmar surface (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - chest & palms of hands (Skin and subcutaneous tissue disorders) | 1 (1)
Rash - soles (Skin and subcutaneous tissue disorders) | 1 (1)
Right hip - slightly limited range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Rigors (General disorders) | 1 (1)
Sacro-iliac pain, right side (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensitive teeth (Gastrointestinal disorders) | 1 (1)
Severe fatigue (General disorders) | 1 (1)
Skin fibrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleepiness (General disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 6 (6)
Stomatitis, candida (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3)
Tachypnea (Cardiac disorders) | 1 (1)
Tearing (Eye disorders) | 2 (2)
Tenderness (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombophlebitis, superficial, B/L (Vascular disorders) | 1 (1)
Total bilirubin, high (Metabolism and nutrition disorders) | 5 (5)
Transfusion, RBC (Blood and lymphatic system disorders) | 2 (2)
Ulceration on right buccal mucosa (Gastrointestinal disorders) | 1 (1)
Vaginal irritation (Reproductive system and breast disorders) | 1 (1)
Vascular: thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Visual changes (Eye disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Allergy/Immunology: Allergic rhinitis (Immune system disorders) | 2 (8)
Ankle edema B/L (Blood and lymphatic system disorders) | 1 (1)
Ankle swelling, bilaterally (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Auditory/Ear: Hearing (Ear and labyrinth disorders) | 1 (3)
Auditory/Hearing: External auditory canal (Ear and labyrinth disorders) | 1 (1)
Blood/Bone Marrow:CD4 Count (Blood and lymphatic system disorders) | 1 (4)
Blood/Bone Marrow:Haptoglobin (Blood and lymphatic system disorders) | 1 (5)
BMT Complex/Multicomponent Events: Graft versus host disease (General disorders) | 1 (2)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1)
C. difficile colitis (Gastrointestinal disorders) | 1 (1)
Cardiac Arrhythmia - Prolonged QTc interval (Cardiac disorders) | 2 (7)
Cardiac Arrhythmia: Supraventricular and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 1 (1)
Cardiac Arrhythmia: Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 2 (4)
Cardiac General: Other, capillary leak syndrome (Cardiac disorders) | 1 (5)
Cardiac General: Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Cardiovascular (Arrhythmia): Sinus bradycardia (Cardiac disorders) | 1 (1)
Cardiovascular General: Cardiac left ventricular function (Cardiac disorders) | 1 (2)
Cardiovascular/General: Other (Specify, venous valve) (Cardiac disorders) | 1 (3)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholesterol (Metabolism and nutrition disorders) | 1 (1)
Coagulation: Other (Specify, bruising to lower extremities) (Blood and lymphatic system disorders) | 1 (1)
Coagulation: INR (International Normalized Ration of prothrombin time) (Blood and lymphatic system disorders) | 7 (29)
Coagulation: Other (Specify, positive lupus anticoagulant) (Blood and lymphatic system disorders) | 1 (1)
Coagulation: thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (3)
Constitutional Symptoms: Rigors/Chills (General disorders) | 4 (5)
Constitutional Symptoms: Sweating (diaphoresis) (General disorders) | 3 (6)
Constitutional Symptoms: Weight gain (General disorders) | 2 (8)
Cystitis (Renal and urinary disorders) | 1 (1)
Death: Death not associated with CTCAE term: Disease progression NOS (General disorders) | 4 (4)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dermatology/Skin: Bruising (Skin and subcutaneous tissue disorders) | 2 (12)
Dermatology/Skin: Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (3)
Dermatology/Skin: Chelitis (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatology/Skin: Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11 (47)
Dermatology/Skin: Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin: Other (Skin and subcutaneous tissue disorders) | 1 (3)
Dermatology/Skin: Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin: Pruritis/itching (Skin and subcutaneous tissue disorders) | 4 (9)
Dermatology/Skin: Radiation dermatitis (Skin and subcutaneous tissue disorders) | 1 (7)
Dermatology/Skin: Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 (24)
Dermatology/Skin: Rash: dermatitis (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatology/Skin: Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (6)
Dermatology/Skin: Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin: Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatology/Skin: Bruising (in absence of Grade 3 (Skin and subcutaneous tissue disorders) | 1 (3)
Dermatology: Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Endocrine: Hot flashes/Flushes (Endocrine disorders) | 1 (1)
Flexion contracture, left knee (musculoskeletal, other) (Musculoskeletal and connective tissue disorders) | 1 (1)
Endocrine: Other (Specify, secondary ovarian failure) (Endocrine disorders) | 1 (1)
Gastrointestinal: Other (Specify, early satiety) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal: Distention/bloating (Gastrointestinal disorders) | 1 (2)
Gastrointestinal: Mucositis/stomatitis - Oral cavity (Gastrointestinal disorders) | 1 (1)
Gastrointestinal: Ascites (non-malignant) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal: Dehydration (Gastrointestinal disorders) | 3 (3)
Gastrointestinal: Colitis (Gastrointestinal disorders) | 3 (4)
Gastrointestinal: (Gastrointestinal disorders) | 2 (4) — Diarrhea associated with graft versus host disease (GVHD) for BMT studies, if specified in the protocol.
Gastrointestinal: Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3 (5)
Gastrointestinal: Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal: Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 (4)
Gastrointestinal: Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 2 (9)
Gastrointestinal: Other (Gastrointestinal disorders) | 1 (1)
Gastrointestinal:other, specify::Cholestasis (Gastrointestinal disorders) | 1 (3)
Gastrointestinal: Proctitis (Gastrointestinal disorders) | 2 (3)
Gastrointestinal: Vomiting (Gastrointestinal disorders) | 5 (8)
Gastrointestinal: Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal: Anorexia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal: Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal: Dehydration (Gastrointestinal disorders) | 1 (1)
Gastrointestinal: Dental:Teeth (Gastrointestinal disorders) | 1 (4)
Gastrointestinal: Nausea (Gastrointestinal disorders) | 2 (2)
Hematochezia/rectal bleeding (Gastrointestinal disorders) | 1 (1)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage/Bleeding: Hematoma (Blood and lymphatic system disorders) | 1 (5)
Hemorrhage/Bleeding: Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 2 (8)
Hemorrhage/Bleeding: Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage/Bleeding: Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (2)
Hemorrhage::Rectal bleeding/hematochezia (Blood and lymphatic system disorders) | 2 (5)
Hemorrhage: Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Hepatic: Albumin, serum-low (hypoalbuminemia) (Hepatobiliary disorders) | 2 (4)
Hepatic:Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 1 (4)
Hepatobiliary/Pancreas:: Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary/Pancreas:: Pancreatitis (Hepatobiliary disorders) | 1 (3)
Increased perirectal pain (Gastrointestinal disorders) | 1 (1)
Infection: Other (Infections and infestations) | 2 (4)
Infection - Other (Specify, abrasion right great toe) (Infections and infestations) | 1 (12)
Infection - Select - Renal/Genitourinary-kidney (Infections and infestations) | 1 (1)
Infection General::Wound (Infections and infestations) | 1 (1)
Infection/Febrile neutropenia::Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with a grade 3 or 4 neutropenia
Infection::Infection (documented clincally or micro) with grade 3 or 4 neutrophils (Infections and infestations) | 3 (3) — (ANC < 1.0x109/l)
Infection::Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2 (3)
Infection::Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically)with Grade 3 or 4 neutrophils (ANC <1.0x10e9/l)::Oral cavity-gums (gingivitis)
Infection::Infection with normal ANC or Grade 1 or 2 neutrophils::Gluteal abscess left side (Infections and infestations) | 1 (1)
Infection::Infection with normal ANC or Grade 1 or 2 neutrophils::Sinusitis (Infections and infestations) | 1 (1)
Infection::Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection::Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 1 (3)
Infection::Opportunistic infection associated with > grade 2 lymphopenia (Infections and infestations) | 1 (6)
Infection::Infection - Other (Specify, clostridium difficile) (Infections and infestations) | 1 (1)
Interstitial nephritis (Renal and urinary disorders) | 1 (1)
Left hip pain/left groin pain (musculoskeletal) (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphatics::Edema:head and neck (Blood and lymphatic system disorders) | 1 (5)
Lymphatics::Lymphatics - Other (Specify, palpable inguinal adenopathy) (Blood and lymphatic system disorders) | 1 (2)
Lymphedema, left LE (Blood and lymphatic system disorders) | 1 (1)
Metabolic/Laboratory: Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13 (195)
Metabolic/Laboratory: Other, (Specify, BUN, high) (Metabolism and nutrition disorders) | 3 (6)
Metabolic/Laboratory: Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (3)
Metabolic/Laboratory: ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 11 (209)
Metabolic/Laboratory: Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 (7)
Metabolic/Laboratory: Creatinine (Metabolism and nutrition disorders) | 5 (17)
Metabolic/Laboratory: Hemogloginuria (Metabolism and nutrition disorders) | 1 (1)
Metabolic/Laboratory: Metabolic/Laboratory: Other, (Specify, LDH) (Metabolism and nutrition disorders) | 20 (163)
Metabolic/Laboratory: Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (32)
Metabolic/Laboratory:Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 11 (102)
Metabolic/Laboratory: Proteinuria (Metabolism and nutrition disorders) | 7 (42)
Metabolic/Laboratory: Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 6 (12)
Metabolic/Laboratory: Other, urine protein (Metabolism and nutrition disorders) | 3 (12)
Mild erythema (IV access site) (Skin and subcutaneous tissue disorders) | 1 (1)
Mild fatigue (General disorders) | 1 (2)
Mucositis of throat and rectal area (Gastrointestinal disorders) | 1 (1)
Mult. abdominal ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Musculoskeletal/Soft tissue: Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft tissue: Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal/Soft tissue: Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft tissue: Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft tissue: Muscular/Skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 1 (6)
Neurology: Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Neurology:Ataxia (incoordination) (Nervous system disorders) | 1 (5)
Neurology: Confusion (Nervous system disorders) | 1 (1)
Neurology: Insomnia (Nervous system disorders) | 1 (3)
Neurology: neuropathy: motor (Nervous system disorders) | 1 (5)
Neurology: other (Nervous system disorders) | 1 (4)
Ocular/Visual:Dry eyes (Eye disorders) | 1 (2)
Pain - Other (Specify, pain at site of biopsy) (General disorders) | 1 (1)
Pain - Other: Breathing (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pain - right lateral (General disorders) | 1 (1)
Pain - Select: Renal/Genitourinary - Kidney (Renal and urinary disorders) | 1 (2)
Pain - Other (General disorders) | 1 (1)
Pain with defecation (Gastrointestinal disorders) | 1 (1)
Pain/Dermatology/Skin::Face (Skin and subcutaneous tissue disorders) | 1 (1)
Pain/Dermatology/Skin::Oral (Skin and subcutaneous tissue disorders) | 1 (1)
Pain/Gastrointestinal::Abdomen NOS (Gastrointestinal disorders) | 9 (39)
Pain/General::Tumor pain (General disorders) | 1 (4)
Pain/Musculoskeletal::Extremity-limb, upper (Musculoskeletal and connective tissue disorders) | 1 (3)
Musculoskeletal::Muscle (Musculoskeletal and connective tissue disorders) | 4 (22)
Pain/Musculoskeletal::Oral cavity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain/Myalgia (Muscle pain) (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain/Neurology::Neuralgia/peripheral nerve (Nervous system disorders) | 1 (2)
Pain/Pulmonary/Upper Respiratory::Throat/pharynx/Larynx (Respiratory, thoracic and mediastinal disorders) | 5 (18)
Pain/Sexual/Reproductive Function::Urethra (Reproductive system and breast disorders) | 1 (2)
Pain:Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain:Earache (Ear and labyrinth disorders) | 1 (1)
Pain:General (General disorders) | 1 (1)
Pain:Musculoskeletal - Joint (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain:Other back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Other hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Other leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Other neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Other upper right quadrant (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Pelvis (Reproductive system and breast disorders) | 1 (1)
Pain:Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pain:Dermatology/Skin - Oral gums (Skin and subcutaneous tissue disorders) | 1 (1)
Pain: Gastrointestinal - Anus (Gastrointestinal disorders) | 2 (3)
Pain::General - Tumor pain (General disorders) | 1 (1)
Pain::Pain - Other (Specify, surgical incision pain) (Injury, poisoning and procedural complications) | 1 (3)
Pain::Pain - Select: Sexual/Reproductive Function - Scrotum (Reproductive system and breast disorders) | 1 (8)
Pain::Pain:: Abdomen NOS (Gastrointestinal disorders) | 1 (3)
Pain::Pain::Back (Musculoskeletal and connective tissue disorders) | 5 (12)
Pain::Pain::Bone (Musculoskeletal and connective tissue disorders) | 5 (17)
Pain::Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain::Pain::Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain::Pain::Head/headache (Nervous system disorders) | 3 (8)
Pain::Pain::Muscle (Musculoskeletal and connective tissue disorders) | 5 (15)
Pain::Pain::Oral cavity (Gastrointestinal disorders) | 2 (5)
Pain::Pain::Paraspinal (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain::Pain::Throat/pharynx/larynx (Gastrointestinal disorders) | 1 (3)
Pain::Head/headache (Nervous system disorders) | 1 (1)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Rectal or perirectal pain (Proctalgia) (Gastrointestinal disorders) | 1 (1)
Perirectal pain (Gastrointestinal disorders) | 1 (1)
Proctitis/perirectal skin breakdown (Gastrointestinal disorders) | 1 (1)
Pulmonary/Upper Respiratory::Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Pulmonary/Upper Respiratory: Cough (Respiratory, thoracic and mediastinal disorders) | 18 (40)
Pulmonary/Upper Respiratory:Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Pulmonary/Upper Respiratory: Fev1 (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pulmonary/Upper Respiratory: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary/Upper Respiratory: Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pulmonary/Upper Respiratory:pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pulmonary/Upper Respiratory: Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pulmonary/Upper Respiratory: Pulmonary/Upper Respiratory: Other (Specify, crackles) (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pulmonary: Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Pulmonary:Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Radiodermatitis, right lateral leg (Skin and subcutaneous tissue disorders) | 1 (3)
Renal/Genitourinary::Dysuria (Renal and urinary disorders) | 2 (2)
Renal/Genitourinary::Obstruction, GU::Ureter (Renal and urinary disorders) | 1 (3)
Renal/Genitourinary::Stricture/Stenosis, GU - Select, left hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary::Urinary frequency/urgency (Renal and urinary disorders) | 1 (2)
Renal/Genitourinary::Urinary retention (Renal and urinary disorders) | 1 (1)
Rhinorrhea (Immune system disorders) | 1 (1)
Sexual/Reproductive Function - Erectile dysfunction (Reproductive system and breast disorders) | 2 (9)
Sexual/Reproductive::Other (Reproductive system and breast disorders) | 1 (3)
Sore rib cage on left side (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Ulcerations - soft palate (Gastrointestinal disorders) | 1 (1)
URI/Sinusitis (Renal and urinary disorders) | 1 (1)
Vascular::Vessel injury - vein-Select:Other NOS (Vascular disorders) | 1 (4)
Verrucae (Skin and subcutaneous tissue disorders) | 1 (1)
Low grade fevers (General disorders) | 1 (1)
Pulmonary emboli, B/L (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection: General, catheter related (Infections and infestations) | 1 (1)
Death (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No